Insert Header with institution's name or institution's letterhead

# **Participant Information Sheet/Consent Form**

Interventional Study - Adult providing own consent Participants receiving SARS-CoV-2 vaccination

[Insert site name]

Title

**Short Title** 

Protocol Number Project Sponsor

Coordinating Principal Investigator/ Principal Investigator

Associate Investigator(s)

Does repeated influenza vaccination constrain influenza immune responses and protection?

**HCW Cohort Study** 



Melbourne Health





**Location** [insert name of hospital].

Thank you for taking the time to read this Information Statement and Consent form. This document is 8 pages long. Please make sure you have all the pages.

# Part 1: What does my participation involve?

#### 1 Introduction

You are invited to take part in this research project because you work at [insert name of hospital]. This is a sub-study of the project 'Does repeated influenza vaccination constrain influenza immune responses and protection?' and will examine the immune response to SARS-CoV-2 vaccination among hospital workers.

This Participant Information Sheet/Consent Form tells you about the research project. It explains the tests involved. Knowing what is involved will help you decide if you want to take part in the research.

Please read this information carefully. Ask questions about anything that you don't understand or want to know more about. Before deciding whether or not to take part, you might want to talk about it with a relative, friend or your local doctor. Participation in this research is voluntary. If you don't wish to take part, you don't have to.

If you decide you want to take part in the research project, you will be asked to sign the consent section. By signing it you are telling us that you:

- Understand what you have read
- Consent to take part in the research project

- Consent to have the tests that are described
- Consent to the use of your personal and health information as described
- Consent to storage and use of samples for future related research

You will be given a copy of this Participant Information and Consent Form to keep.

## 2 What is the purpose of this research?

The purpose of this project is to examine the immune response to SARS-CoV-2 (the virus that causes COVID-19 disease) vaccination among hospital staff by measuring antibody levels.

People who are vaccinated against SARS-CoV-2 develop antibodies which protect against the virus. When a vaccinated person is exposed to SARS-CoV-2, these antibodies latch onto the virus and remove it from the body.

As SARS-CoV-2 vaccines are new, more studies are required to understand the immune response to the different vaccines, as well as whether the order of SARS-CoV-2 and influenza vaccinations matters. The findings from this sub-study may provide information contributing to this area of research.

#### 3 What does participation in this research involve?

This research project is a sub-study of the influenza study and consists of a main sub-study and nested sub-study. If you agree to participate you will be enrolled into either the main sub-study or the nested sub-study.

The total time commitment for participating in this sub-study is approximately 4 hours per year for [insert number of years depending on year of enrolment] years.

There are no costs associated with your participation in this research project, nor will you be paid. All tests required as part of the research project will be provided to you free of charge. Each time you are seen for a blood sample, you will be given

# 3.4 Main sub-study

Participation in the main sub-study will involve at least one additional blood sample collected 14-21 days after the completed course of the SARS-CoV-2 vaccine (commonly after the 2<sup>nd</sup> dose). If the study does not have a pre-SARS-CoV-2 vaccination blood sample for your already, you will also be asked to provide a SARS-CoV-2 pre-vaccination sample. The schedule for collection of blood samples is as follows:



#### 3.5 Nested sub-study

Participation in the nested sub-study will involve 2-3 additional blood samples for sera, as well as PBMC and plasma. These will be collected at 7 and 14-21 days after the completed course of SARS-CoV-2 vaccine (commonly after the 2<sup>nd</sup> dose). If the study does not have a pre-SARS-CoV-2 vaccination blood sample for you already, you will also be asked to provide a SARS-CoV-2 pre-vaccination sample. The schedule for collection of blood samples is as follows:



#### 4 What do I have to do?

To participate in this sub-study, you must be:

- enrolled in the associated influenza study
- aged between 18 and 60 years;
- a current staff, student, volunteer or honorary member at [insert hospital name] eligible for the hospital's free vaccination program;
- willing to provide a current mobile phone number for SMS reminders during the study period
- have a mobile phone that can receive and send SMS messages;
- able and willing to complete the informed consent process;
- able and willing to provide follow up blood samples;
- available for follow-up over the next 7 months.

You will not be able to participate in this sub-study if you have received immunosuppressive treatment within the past 6 months or are contraindicated for SARS-CoV-2 vaccine

#### 5 Other relevant information about the research project

Six hospitals in Australia will participate in this study. [Insert hospital name] is one of the participating hospitals. A total of 250 staff at [insert hospital name] will participate in the influenza study. Overall, 1500 healthcare workers across 6 hospitals will participate in the study.

This research has been funded by the US National Institutes of Health

#### 6 Do I have to take part in this research project?

Participation in any research project is voluntary. If you do not wish to take part, you do not have to. If you decide to take part and later change your mind, you are free to withdraw from the project at any stage. If you do decide to take part, you will be given this Participant Information and Consent Form to sign and you will be given a copy to keep. Your decision whether to take part or not to take part, or to take part and then withdraw, will not affect your relationship with [insert hospital name].

## 7 What are the alternatives to participation?

You do not have to take part in this research project. This is a research study and does not constitute treatment or therapy.

## 8 What are the possible benefits of taking part?

We cannot guarantee or promise that you will receive any benefits from this sub-study. This study may be able to provide previously unknown information about SARS-CoV-2 antibody levels in hospital workers. This information is useful for vaccination programmes in hospitals. This information is useful for SARS-CoV-2 vaccination programmes in hospitals. You will be able to find out how well your body has responded to vaccination using one measure of antibody response.

#### 9 What are the possible risks and disadvantages of taking part?

Blood samples will be collected as part of the sub-study. There are no major risks associated with giving blood. Most people feel uncomfortable when the needle is put in their arm to take blood. It is possible there may be some bruising, swelling, or bleeding where the needle enters the skin.

# 10 What will happen to my test samples?



## 11 What if new information arises during this research project?

Sometimes during the course of a research project, new information about the risks and benefits of the project may become available. If this happens, the study coordinator will tell you about it and discuss with you whether you want to continue in the research project. If you decide to withdraw you will be free to do so at this time. If you decide to continue in the research project you will be asked to sign an updated consent form.

## 12 What if I withdraw from this research project?

If you decide to withdraw from the project, please notify a member of the research team before you withdraw. This notice will ensure the study team do no try to contact you for follow-up. If you do withdraw your consent during the research project, the research team will not collect additional personal information from you, although personal information already collected will be retained to ensure that the results of the research project can be measured properly and to comply with law.

# Part 2: How is the research project being conducted?

#### 13 What will happen to information about me?

By signing the consent form you consent to the study doctor and relevant research staff collecting and using personal information about you for the research project. Any information obtained for the purpose of this research project that can identify you will be treated as confidential and securely stored. It will be disclosed only with your permission, or as required by law.

Additional information on vaccine brand and batch numbers will be collected from [insert name of department that holds vaccination records]. The study data will be collected, stored and archived together with your original consent form in

It is anticipated that the results of this research project will be published and/or presented in a variety of forums. In any publication and/or presentation, information will be provided in such a way that you cannot be identified. You will be able to obtain a copy of any publications from the study website [insert url].

In accordance with relevant Australian and/or Victorian privacy and other relevant laws, you have the right to request access to your information collected and stored by the research team. You also have the

right to request that any information with which you disagree be corrected. Please contact the study team member named at the end of this document if you would like to access your information.

## 14 Complaints and compensation

If you suffer any injuries or complications as a result of this research project, you should contact the study team as soon as possible and you will be assisted with arranging appropriate medical treatment. If you are eligible for Medicare, you can receive any medical treatment required to treat the injury or complication, free of charge, as a public patient in any Australian public hospital.

#### 15 Who is organising and funding the research?

This research project is being conducted by , in collaboration with [enter department and hospital name]. The research project is funded by the US National Institutes of Health. No member of the research team will receive a personal financial benefit from your involvement in this research project (other than their ordinary wages).

#### 16 Who has reviewed the research project?

All research in Australia involving humans is reviewed by an independent group of people called a Human Research Ethics Committee (HREC). The ethical aspects of this research project have been approved by the HREC of Melbourne Health.

This project will be carried out according to the *National Statement on Ethical Conduct in Human Research* (2007). This statement has been developed to protect the interests of people who agree to participate in human research studies.

#### 17 Further information and who to contact

The person you may need to contact will depend on the nature of your query. If you want any further information concerning this project or if you have any medical problems which may be related to your involvement in the project (for example, any side effects), you can contact the coordinating principal investigator or any of the following people:

## **Study coordinator**

| Name | [Name] |
|-----------|-----------------|
| Position | [Position] |
| Telephone | [Phone number] |
| Email | [Email address] |

#### Clinical contact person

| | policion. |
|-----------|-----------------|
| Name | [Name] |
| Position | [Position] |
| Telephone | [Phone number] |
| Email | [Email address] |

For matters relating to research at the site at which you are participating, the details of the local site complaints person are:

#### **Complaints contact person**

| Name | [Name] |
|-----------|-----------------|
| Position | [Position] |
| Telephone | [Phone number] |
| Email | [Email address] |

If you have any complaints about any aspect of the project, the way it is being conducted or any questions about being a research participant in general, then you may contact:

| Reviewing HREC name | Melbourne Health |
|------------------------|------------------|
| HREC Executive Officer | |

| Telephone |
|-----------|
| Email |

# Reviewing HREC approving this research and HREC Executive Officer details

# **Local HREC Office contact (Single Site - Research Governance Officer)**

| Name | [Name] |
|-----------|-----------------|
| Position | [Position] |
| Telephone | [Phone number] |
| Email | [Email address] |

# **Consent Form -** Adult providing own consent

| Title | Does repeated influenza vaccination constrain influenza immune responses and protection? |
|---|---|
| Short Title | HCW Cohort Study |
| Protocol Number | The William Study |
| | Naula avena a Lla altila |
| Project Sponsor | Melbourne Health |
| Coordinating Principal Investigator/<br>Principal Investigator | |
| Associate Investigator(s) (if required by institution) | |
| Location (where CPI/PI will recruit) | [Location where the research will be conducted] |
| understand. I understand the purposes, procedure I have had an opportunity to ask quest I freely agree to participate in this rese withdraw at any time during the study I understand that I will be given a sign. I will be participating in (the sub-study Study Doctor/Senior Researcher befor Main SARS-CoV-2 vaccination some Nested SARS-CoV-2 vaccination Declaration by Participant – for participan | vallocation information below was provided to me by the re signing this consent form): ub-study sub-study nts who have read the information |
| Signature | Date |
| Witness to the informed consent process Name (please print) Signature * Witness is not to be the investigator, a member the interpreter may not act as a witness to the con Declaration by Study Doctor/Senior Research I have given a verbal explanation of the reparticipant has understood that explanation Name of Study Doctor/ | ice CPMP/ICH/135/95 Section 4.8.9, witness * required Date of the study team or their delegate. In the event that an interpreter is used, essent process. Witness must be 18 years or older. archer† search project, its procedures and risks and I believe that the |
| Senior Researcher <sup>†</sup> (please print) | |

Master Participant Information Sheet/Consent Form 22 March 2021 (Complete if required) [Site Name] Site Master Participant Information Sheet/Consent Form [Date] Local governance version [Date] (Site PI use only)

| Signature Date |
|---|
| <sup>†</sup> A senior member of the research team must provide the explanation of, and information concerning, the research project.<br>Note: All parties signing the consent section must date their own signature. |
| Consent to use of samples for future research |
| I consent to the storage and use of blood and swabs taken from me for use, as described in the relevant section of the Participant Information Sheet, for (please check all that apply): This specific research project Other research that is closely related to this research project Any future research. |
| Name of Participant (please print) |
| Signature Date |
| For participants <u>unable</u> to read the information and consent form |
| See Note for Guidance on Good Clinical Practice CPMP/ICH/135/95 Section 4.8.9, witness * required Witness to the informed consent process Name (please print) |
| Signature Date |
| * Witness is <u>not</u> to be the investigator, a member of the study team or their delegate. In the event that an interpreter is used, the interpreter may <u>not</u> act as a witness to the consent process. Witness must be 18 years or older. |
| Name of Study Doctor/ Senior Researcher <sup>†</sup> (please print) |
| Signature Date |

<sup>&</sup>lt;sup>†</sup> A senior member of the research team must provide the explanation of and information concerning the research project. Note: All parties signing the consent section must date their own signature.

# Form for Withdrawal of Participation - Adult providing own consent

It is recommended that this form NOT be included as part of the PICF itself, but that it be developed at the same time and made available to researchers for later use, if necessary. Note that a participant's decision to withdraw their separate consent to the use and storage of tissue will need to be documented separately and linked to the PICF used for that purpose.

| Title Short Title Protocol Number Project Sponsor Coordinating Principal Investigator/ Principal Investigator Associate Investigator(s) (if required by institution) | Does repeated influenza vaccination constrain influenza immune responses and protection? HCW Cohort Study Melbourne Health |
|---|---|
| Location (where CPI/PI will recruit) | [Location where the research will be conducted] |
| | e above research project and understand that such ment, my relationship with those treating me or my |
| Signature | Date |
| In the event that the participant's decision to wi<br>Researcher will need to provide a description of | ithdraw is communicated verbally, the Study Doctor/Senior<br>the circumstances below. |
| Declaration by Study Doctor/Senior Resea I have given a verbal explanation of the impedieve that the participant has understood Name of Study Doctor/ | plications of withdrawal from the research project and I |
| Senior Researcher <sup>†</sup> (please print) | |
| Signature | Date |
| <sup>†</sup> A senior member of the research team must provid research project. | e the explanation of and information concerning withdrawal from the |

Master Participant Information Sheet/Consent Form 22 March 2021
(Complete if required) [Site Name] Site Master Participant Information Sheet/Consent Form [Date]
Local governance version [Date] (Site PI use only)

Note: All parties signing the consent section must date their own signature.